CLINICAL TRIAL: NCT07088718
Title: Prediction of the SURPASS-CVOT Cardiovascular Outcome Trial in Healthcare Claims Data
Acronym: DUP-SURPASS
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-SURPASSCVOT
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes; Major Adverse Cardiac Events; Cardiovascular (CV) Risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Tirzepatide; dulaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tirzepatide: Exposure group
  Interventions: Drug: Tirzepatide
- Dulaglutide: Reference group
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Tirzepatide — New use of tirzepatide dispensing claim is used as the exposure.
  Groups: Tirzepatide
Drug: Dulaglutide — New use of dulaglutide dispensing claim is used as the reference.
  Groups: Dulaglutide

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale emulation of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the Randomized Controlled Trials Duplicated Using Prospective Longitudinal Insurance Claims: Applying Techniques of Epidemiology (RCT-DUPLICATE) initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to emulate, as closely as is possible in healthcare insurance claims data, the SURPASS-CVOT trial described below. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization cannot be achieved in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides guidance on the reference standard treatment effect estimate. However, failure to replicate RCT findings is not necessarily indicative of the inadequacy of the healthcare claims data for emulation for a range of possible reasons and does not provide information on the validity of the original RCT finding.

The SURPASS-CVOT trial is a non-inferiority trial that aims to evaluate the effect of tirzepatide, a dual glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide-1 receptor agonist (GLP-1-RA), vs dulaglutide, a GLP-1-RA, on time to first occurrence of any major adverse cardiovascular event (MACE), defined as cardiovascular death, myocardial infarction, or stroke among patients with type 2 diabetes mellitus (T2DM) and an established cardiovascular disease (CVD). In addition, the trial aims to determine noninferiority with a magnitude of difference that also supports superiority against putative placebo and for superiority to dulaglutide will be performed. With estimated study completion in summer 2025, results of the trial are yet to be announced. Therefore, we aim to predict the results of the SURPASS-CVOT trial by emulating its design with protocol registration and statistical analysis conducted before the results of the trial are made public.

The database study designed to emulate the SURPASS-CVOT trial will be a new-user active-comparative study, conducted using 2 national United States claims databases, where we compare the effect of tirzepatide vs dulaglutide on the composite end point of all-cause mortality, myocardial infarction, or stroke. Clinical guidelines during the study period recommended both agents under investigation as second-line options for glucose lowering and were similarly costly.

ELIGIBILITY:
FOLLOWING ELIGIBILITY CIRTERIA OF THE SURPASS-CVOT TRIAL

Inclusion Criteria:

* History of MI, surgical or percutaneous coronary/carotid peripheral artery revascularization
* BMI ≥25.0kg/m2
* Type 2 diabetes, diagnosis of coronary/carotid/peripheral artery disease
* Age ≥40 years
* Male or female sex

Exclusion Criteria:

* Medullary thyroid carcinoma, MEN syndrome type 2, malignancy
* Treatment for diabetic retinopathy//macular edema, pancreatitis, gastric emptying abnormality/bariatric surgery, liver disease, end-stage renal disease or dialysis, pregnancy
* Prior use of pramlintide or any GLP-1-RA except tirzepatide or dulaglutide
* Cardiovascular event, hospitalization for heart failure
* Concurrent use of both drugs i.e. tirzepatide and dulaglutide

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 40 years or older with T2DM and an established CVD
Sampling Method: Non-Probability Sample
Enrollment: 44671 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
First occurence of MACE (all-cause mortailty, myocardial infarction, or death) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs dulaglutide on time to first occurrence of MACE (all-cause mortailty, myocardial infarction, or death) in patients with T2DM and an established CVD when following the eligibility criteria of the SURPASS-CVOT trial: Individuals aged 40 years or older with T2DM and an established CVD.

SECONDARY OUTCOMES:
Individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke (Tirzepatide vs dulaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs dulaglutide on the individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke in patients with T2DM and an established CVD when following the eligibility criteria of the SURPASS-CVOT trial: Individuals aged 40 years or older with T2DM and an established CVD.
Hernia | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the effect of tirzepatide vs dulaglutide on a negative control outcome of hernia in patients with T2DM and an established CVD when following the eligibility criteria of the SURPASS-CVOT trial: Individuals aged 40 years or older with T2DM and an established CVD.
Lumbar radiculopathy | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the effect of tirzepatide vs dulaglutide on a negative control outcome of lumbar radiculopathy in patients with T2DM and an established CVD when following the eligibility criteria of the SURPASS-CVOT trial: Individuals aged 40 years or older with T2DM and an established CVD.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital; Nils Krüger, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kruger N, Schneeweiss S, Desai RJ, Sreedhara SK, Kehoe AR, Fuse K, Hahn G, Schunkert H, Wang SV. Cardiovascular outcomes of semaglutide and tirzepatide for patients with type 2 diabetes in clinical practice. Nat Med. 2025 Nov 9. doi: 10.1038/s41591-025-04102-x. Online ahead of print. PMID 41207920

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Amendment 1 to Study Protocol and Statistical Analysis Plan (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT07088718/Prot_SAP_002.pdf
  • Study Protocol and Informed Consent Form: Study Protocol and Statistical Analysis Plan (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT07088718/Prot_ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan: Amendment 2 to Study Protocol and Statistical Analysis Plan (2025-10-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT07088718/Prot_SAP_003.pdf